CLINICAL TRIAL: NCT05960331
Title: Influence of Autonomy on Motor Learning in People With Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202304047RINC
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Autonomy; Motor learning; Transcranial magnetic stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-control group (Experimental): Participants will be able to choose over feedback schedule when practicing finger-pressing trajectory matching task.
  Interventions: Behavioral: Autonomy supported learning
- Yoked group (Active Comparator): Participants will receive feedback, which was determined by their counterpart in self-control group, with no-choice when practicing finger-pressing trajectory matching task.
  Interventions: Behavioral: Practice with predetermined feedback

INTERVENTIONS:
Behavioral: Autonomy supported learning — The ability of learners to participate in determining their own behaviour, which is the feedback schedule regarding their practice performance in this study.
  Arms: Self-control group
Behavioral: Practice with predetermined feedback — Learners practice the motor task, while the feedback is provided according to their counterpartner
  Arms: Yoked group

SUMMARY:
The goal of this clinical trial is to explore the benefits of autonomy supported learning in patients with Parkinson's disease. The main questions to answer are:

* Whether autonomy supported learning can benefit motor learning in PD patients
* Whether autonomy supported learning can enhance intrinsic motivation and/ or information processing of PD patients in learning a new task.
* Whether autonomy supported learning can facilitate cortical excitability change after practicing a new task.

Participants will be recruited into two groups (Self-control group, SC; and yoked group, YK) to learn a finger-pressing trajectory matching task

* Participants in SC group will have choice over feedback schedule during trial practice
* Participants in YK group will receive feedback with no-choice during trial practice Researchers will compare the retention test performance to see if autonomy supported learning will lead to better learning effect.

DETAILED DESCRIPTION:
Autonomy is the sense of learner to actively participate in determining their own behaviour. The present study aims to investigate whether an autonomy supported practice (with self-controlled feedback) would benefit adults with Parkinson's disease (PD), along with increased intrinsic motivation, information processing and cortical excitability. Two groups of healthy adults and two groups of PD patients will be recruited to learn a finger-pressing trajectory matching task. Participants will be allocated in either a self-control group (choice over feedback schedule), or a yoked group (receive feedback with no-choice). Learning will be assessed on the second day and one week later, along with an error estimation of learners' own performance to represent their information processing ability. Cortical excitability and inhibition will be assessed via transcranial magnetic stimulation as indicators of cortical plasticity. Questionnaire regarding motivation will be assessed before and after practice trials. Study hypothesized that individual with PD would benefit from autonomy supported learning, with better performance, enhanced motivation and information processing, associates with change of cortical excitability

ELIGIBILITY:
Inclusion Criteria:

* age above 20-years-old
* able to follow instructions to perform the tasks (Montreal Cognitive Assessment ≥ 24)
* no surgery and injury in upper extremities in recent 6 months

Exclusion Criteria:

* other neurological disorders in addition to Parkinson's disease
* Parkinson's disease dementia
* symptom of severe tremor in upper extremities (score ≥ 3 in Question 15 to 18 of UPDRS-III)
* deep brain stimulation or pacemaker implanted
* medical history of seizure
* a blood-relative with history of epilepsy
* unstable medical conditions
* pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Performance accuracy | up to day 7
  Overall performance accuracy relative to the target waveform was assessed using root mean square error (RMSE), which is the mean difference between the target waveform and the participant's movement trajectory calculated over their actual movement time.

SECONDARY OUTCOMES:
Intrinsic Motivation Inventory | day 1, day 2, day 7
  A questionnaire with subscales of perceived competence and autonomy. Questions were either taken directly or modified from the IMI, regarding to the participants subjective motivation after completing their practice trials.
Error Estimation | day 2, day 7
  Participants will be instructed to estimate their error in RMSE after completing each trial in retention and transfer test. Error estimation is used to assess the cognitive processing of participants during the trials.
Cortical excitability changes | Baseline, day 2, day 7
  Transcranial magnetic stimulation (TMS) device (The Magstim Company Ltd, Whitland, UK) will be used to determine the neurophysiological changes of corticomotor excitability before and after the acquisition phase.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carter MJ, Ste-Marie DM. Not all choices are created equal: Task-relevant choices enhance motor learning compared to task-irrelevant choices. Psychon Bull Rev. 2017 Dec;24(6):1879-1888. doi: 10.3758/s13423-017-1250-7. PMID 28224481
- [Result] Chiviacowsky S, Wulf G, Lewthwaite R, Campos T. Motor learning benefits of self-controlled practice in persons with Parkinson's disease. Gait Posture. 2012 Apr;35(4):601-5. doi: 10.1016/j.gaitpost.2011.12.003. Epub 2011 Dec 30. PMID 22209649